CLINICAL TRIAL: NCT03158337
Title: Effects of Regular Exercise on Cerebrovascular Reserve in Older Adults: Role in the Prevention of Age-Related Cognitive Decline
Brief Title: Effects of Regular Exercise on Cerebrovascular Reserve in Older Adults
Acronym: BIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Marc Poulin, Professor, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: E-22502
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Aging; Physical Activity; Cognitive Function
Keywords: Exercise; Physical Activity; Brain blood flow; Cognition; Fitness
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aerobic exercise (Experimental): Participants took part in a supervised 6-month long aerobic (walk/jog) training program held 3 days/week. Each session included a 5-min warm-up, 20-40 min of aerobic exercise (walking, jogging), 5-min cool-down, and stretching. Exercise prescriptions follow current principles and guidelines established by ACSM/AHA, including sufficient warm-up, cooldown, and ongoing provision of safety precautions/exercise tips. As participants progress, the duration of aerobic exercise increased from 20 (month 1) to 30 (months 2-3) and 40 min (months 4-6), with proportional increases to warm-up and cool-down periods. Exercise intensity is based on individual maximal oxygen uptake (VO2 max), measured at baseline. Intensity builds from 30-45% (months 1-3) to mitigate the risk of injury and will progress to 60-70% (months 4-6) heart rate reserve (HRR).
  Interventions: Behavioral: Aerobic exercise

INTERVENTIONS:
Behavioral: Aerobic exercise

SUMMARY:
While it is well established that physical inactivity is a modifiable risk factor for vascular disease and cognitive decline, the mechanism by which exercise exerts its protective effect on the cerebral circulation and cognition is unknown. This knowledge gap was recognized recently in the Centers for Disease Control & Prevention and the Alzheimer's Association document "National Public Health Road Map to Maintaining Cognitive Health". Our rationale for these studies is that the identification of physical exercise as a lifestyle factor able to improve cerebrovascular reserve and cognition would establish a strong scientific framework justifying design of a randomized clinical trial that could evaluate the role of physical activity in cerebrovascular health and function.

This research is based on data we obtained from a cross-sectional study that showed significant relations between physical fitness, vascular regulation and cognition. Cerebrovascular reserve and cognition were better maintained in women who were physically active but reduced in women who were sedentary. Our central hypothesis is that regular aerobic exercise mitigates age-related decreases in cerebrovascular reserve, which in turn imparts benefits in cognition. Further, we believe that these effects will persist after the structured aerobic exercise program is terminated.

Our 18 month study began with a 6-month baseline period, followed by a 6-month exercise intervention, and a 6-month follow-up period. In addition, there are 5-year and 10-year follow-up periods. Volunteers (men and women aged ≥ 55 years) from the community were recruited using a variety of recruitment methods including media and distribution lists. After the baseline (pre-training) measurements, participants underwent a six-month aerobic training program, following guidelines previously used by us and according to the new exercise guidelines for older adults established by American College of Sports Medicine and the American Heart Association. The study involves comprehensive assessments of physical fitness, cerebrovascular responses to carbon dioxide at rest and during sub-maximal exercise, and an extensive battery of cognitive function tests.

ELIGIBILITY:
Inclusion Criteria:

* sedentary status (engages in less than 30 minutes of moderate exercise four days per week or 20 continuous minutes of vigorous exercise two days per week), the ability to walk independently outside or on stairs, body mass index (BMI) < 35 kg/m^2, women were at least 12 months postmenopausal on entry into the study

Exclusion Criteria:

* heart/chest pain upon physical exertion, fainting spells/dizziness, surgery or major trauma in the previous 6 months, known asthma or sleep apnea, history of myocardial infarction, angina, arrhythmia, valve disease, chronic heart failure, history of stroke, cardiovascular or cerebrovascular disease, history of chronic headache or migraines, history of blood clots/thrombosis, smokers (within last 12 months), currently taking medication (beta-blockers, anti-depressants, digitalis/digoxin, blood thinners (warfarin), evista (raloxifene), corticosteroids (e.g., prednisone), adrenaline/epinephrine, anti-arrhythmics (e.g., norpace)).

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2010-05-01 (Actual); Primary Completion 2016-05-05 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Cognition Assessed by Neuropsychological Test Battery | Measured at baseline (0 and 6 months), exercise intervention completion (12 months) and follow up (18,72 and 132 months)

SECONDARY OUTCOMES:
Change in Maximal Oxygen Uptake (VO2max) Assessed by Metabolic Cart | Measured at baseline (0 and 6 months), during the exercise intervention (9 months), exercise intervention completion (12 months) and follow up (18,72 and 132 months)
Change in Cerebral Blood Flow Assessed by Transcranial Doppler Ultrasound | Measured at baseline (0 and 6 months), during the exercise intervention (9 months), exercise intervention completion (12 months) and follow up (18,72 and 132 months)
Change in Blood Biomarkers Assessed by Elisa Assays | Measured at baseline (0 and 6 months), during the exercise intervention (9 months), exercise intervention completion (12 months) and follow up (18,72 and 132 months)
Change in Risk/protective factors Assessed by Questionnaires | Measured at baseline (0 and 6 months), during the exercise intervention (9 months), exercise intervention completion (12 months) and follow up (18,72 and 132 months)
  Measures include changes in dietary intake, food frequency, supplement intake, physical activity, cognitive activities, mood changes, social support and engagement.

OTHER OUTCOMES:
Change in Sleep Quality Assessed by Polysomnography, Actigraphy and Questionnaires | A sub-sample of participants were assessed at baseline (6 months), exercise intervention completion (12 months) and follow up (18,72 and 132 months).
Change in Brain Structure and Function Assessed by Neuroimaging Modalities | A sub-sample of participants were assessed at baseline (6 months), exercise intervention completion (12 months) and follow up (18,72 and 132 months).

CONTACTS AND LOCATIONS:
Overall Officials: Marc J Poulin, PhD, DPhil, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Background] Tyndall AV, Davenport MH, Wilson BJ, Burek GM, Arsenault-Lapierre G, Haley E, Eskes GA, Friedenreich CM, Hill MD, Hogan DB, Longman RS, Anderson TJ, Leigh R, Smith EE, Poulin MJ. The brain-in-motion study: effect of a 6-month aerobic exercise intervention on cerebrovascular regulation and cognitive function in older adults. BMC Geriatr. 2013 Feb 28;13:21. doi: 10.1186/1471-2318-13-21. PMID 23448504
- [Result] Pannu T, Sharkey S, Burek G, Cretu D, Hill MD, Hogan DB, Poulin MJ. Medication use by middle-aged and older participants of an exercise study: results from the Brain in Motion study. BMC Complement Altern Med. 2017 Feb 10;17(1):105. doi: 10.1186/s12906-017-1595-5. PMID 28187744
- [Result] Gill SJ, Friedenreich CM, Sajobi TT, Longman RS, Drogos LL, Davenport MH, Tyndall AV, Eskes GA, Hogan DB, Hill MD, Parboosingh JS, Wilson BJ, Poulin MJ. Association between Lifetime Physical Activity and Cognitive Functioning in Middle-Aged and Older Community Dwelling Adults: Results from the Brain in Motion Study. J Int Neuropsychol Soc. 2015 Nov;21(10):816-30. doi: 10.1017/S1355617715000880. PMID 26581793
- [Result] Tyndall AV, Argourd L, Sajobi TT, Davenport MH, Forbes SC, Gill SJ, Parboosingh JS, Anderson TJ, Wilson BJ, Smith EE, Hogan DB, Hill MD, Poulin MJ. Cardiometabolic risk factors predict cerebrovascular health in older adults: results from the Brain in Motion study. Physiol Rep. 2016 Apr;4(8):e12733. doi: 10.14814/phy2.12733. PMID 27117804
- [Result] Ishigami Y, Eskes GA, Tyndall AV, Longman RS, Drogos LL, Poulin MJ. The Attention Network Test-Interaction (ANT-I): reliability and validity in healthy older adults. Exp Brain Res. 2016 Mar;234(3):815-27. doi: 10.1007/s00221-015-4493-4. Epub 2015 Dec 8. PMID 26645310
- [Result] Drogos LL, Gill SJ, Tyndall AV, Raneri JK, Parboosingh JS, Naef A, Guild KD, Eskes G, Hanly PJ, Poulin MJ. Evidence of association between sleep quality and APOE epsilon4 in healthy older adults: A pilot study. Neurology. 2016 Oct 25;87(17):1836-1842. doi: 10.1212/WNL.0000000000003255. PMID 27777343